CLINICAL TRIAL: NCT06017440
Title: Effect of Acute Exercise on Sensory and Hedonic Responses to a Fixed Meal in Adolescents With Obesity
Acronym: SMASH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: RBHP 2023 BOIRIE 3; 2023-A00808-37 (Other: ANSM)
Record Dates: First submitted 2023-06-13; First posted 2023-08-30 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: CONTROL Condition; Exercise
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- adolescents with obesity (Experimental): There is only one arm as this is an acute randomized study comparing two differents conditions within the same sample of participants.
  Interventions: Behavioral: EXERCISE; Behavioral: CONTROL

INTERVENTIONS:
Behavioral: EXERCISE — Participants will receive at 08:00 am a calibrated breakfast of 500kcal. They should not perform physical exercise during the day. They will be asked at 11 a.m. to cycle for 30 minutes at 65% of the maximal capacities and their energy expenditure will be measured by indirect calorimetry. At 11 a.m., teenagers will receive a calibrated meal of 800 kcal respecting the nutritional recommendations for this age. Questionnaires on feelings of hunger will be distributed to them at regular intervals. They will also be asked to complete a 10-minute computer exercise to assess their relationship to food before and after lunch (LFPQ. Leeds Food Preference Questionnaire, Liking/ wanting). Finally, from 60 minutes after the midday test meal, teenagers will have access to an ad libitum buffet for one hour.
Behavioral: CONTROL — Teenagers should not perform any physical activity during the day and they will be asked to stay at 11 a.m., for 30 minutes, resting in a semi-supine position.

SUMMARY:
While long considered independently, energy expenditure and energy intake have been shown to interact. Fot the last 20 years, the litterature has been describing tyhe effects of an acute bout of exercise on subsequent energy intake and appetitive responses, indicating a potenital anorexigenic effect of intensive exercise in adolescents with obesity. These studies suggest a decrease in hunger, redcued satiety and modified food reward responses.

These results remain however obtained in studies using post exercise ad libitum test meals and this nature of the meal might ahve impact these responses.

The present work tends to assess the effect of acute exercise on subsequent appetite and food reward responses to a fixed meal, in adolescents with obesity.

DETAILED DESCRIPTION:
After an inclusion visit to ensure the aptitude of adolescents to complete the entire study, each will have to carry out densitometric measurements (body composition and bone structure). The adolescents will then carry out, in a randomized manner, 2 experimental sessions spaced at least 7 days apart: i) a control session (CON); ii) a session with a pedaling exercise at 65% of their estimated maximum capacity (EX).

During each of these experimental sessions, teenagers will receive a calibrated breakfast at 08:00 am. During the CON session, teenagers should not perform any physical activity during the day and they will be asked to stay at 11 a.m., for 30 minutes, resting in a semi-supine position. During the EX session, teenagers will perform moderate-intensity physical exercise (65% of their estimated maximum capacity) at 11 a.m. At noon, the teenagers will have to consume a calibrated meal. Questionnaires on feelings of hunger will be distributed to them at regular intervals. They will also be asked to complete a 10-minute computer exercise to assess their relationship to food just before and just after the calibrated midday meal (LFPQ. Leeds Food Preference Questionnaire, Liking/Wanting, French version). Sixty minutes after the calibrated meal, teenagers will have an ad libitum buffet available for one hour.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 11 to 16 years (inclusive limits), maturation stage 3-5 according to the Tanner classification, with obesity defined by a body mass index (BMI) greater than the 97th percentile according to national curves (Roland- Cachera et al., 1991).
* Adolescent who has signed the information and consent form and whose holders of parental authority have signed the information and consent form
* Person subject to a Social Security scheme

Exclusion Criteria:

Medical or surgical history deemed by the investigator to be incompatible with the study

* Presence of diabetes, and any other pathology limiting the application of one or the other strategy to the trial.
* Taking medications that may interfere with the results of the study
* Subjects with cardiovascular problems, here we are talking about subjects with a history of cardiovascular and/or neurovascular pathology, as well as subjects presenting cardiovascular and/or neurovascular risk factors (excluding obesity/ overweight).
* Surgical intervention in the previous 3 months.
* Subjects undergoing energy restriction or weight loss program through physical activity at the time of inclusion or during the last six months.
* Consumption of tobacco or alcohol.
* Special diet.
* Participation in regular and intense physical and sports activities for more than two hours per week.
* Teenagers whose parents are under guardianship, curatorship, safeguard of justice or not subject to a social security system
* Refusal to sign the information and consent notice
* Person in period of exclusion from another study
* Pregnant or breastfeeding adolescents on declarative

Ages: 11 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 16 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2023-09-17 (Actual); Study Completion 2023-10-17 (Actual)

PRIMARY OUTCOMES:
APPETITE FEELINGS | immediately after lunch
  appetite sensation will be assessed using visual analog scales
FOOD reward | at lunch time
  food reward will be assessed using the leeds food preference questionnaire
Energy intake | at lunch time
  energy intake will be assessed ad libitum at the following diner

CONTACTS AND LOCATIONS:
Overall Officials: Yves Boirie, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, France